CLINICAL TRIAL: NCT04087616
Title: Internet-based -Guided Self-help Intervention for Children With Chronic Tics Syndrome or Tourette Syndrome: Comprehensive Behavioral Intervention for Tics (CBIT) Versus Waiting List: Reduction of Tic Severity and Quality of Life Measures
Brief Title: Internet-based CBIT for Children With Chronic Tics
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tel Aviv Medical Center (Other)
Responsible Party: Principal Investigator, Michael Rotstein, Head, Pediatric Movement Disorder Clinic, Principal Investigator, Tel-Aviv Sourasky Medical Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: TelAvivSMO
Record Dates: First submitted 2019-07-24; First posted 2019-09-12 (Actual); Last update posted 2019-09-12 (Actual); Status verified 2019-09

CONDITIONS: Tourette Syndrome in Children; Tourette Syndrome in Adolescence; Chronic Tic Disorder
Keywords: tics; tourette Syndrome
MeSH Terms: conditions — Tic Disorders; Tics; Tourette Syndrome | interventions — Waiting Lists

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBIT (Experimental): ICBIT. Intervention delivered through an internet platform called Managing children's' tics (www.cbteamathome.co.il), based on CBIT protocol (Woods et al., 2008) adapted to an online parent-guided self-help format.
  Interventions: Behavioral: ICBIT
- Waiting List (Placebo Comparator): Participants initially assigned to the wait list receive no psychosocial intervention for 9 weeks. Following post-WL assessment, all participants receive ICBIT.
  Interventions: Behavioral: waiting list

INTERVENTIONS:
Behavioral: ICBIT — The intervention consists of 9 modules delivered over 9 weeks comprise of age-appropriate texts and descriptive diagrams, animations, films of clinicians demonstrating techniques such as competing response exercising.
  Arms: CBIT
Behavioral: waiting list — Participants initially assigned to the wait list received no psychosocial intervention for 9 weeks. Following post-WL assessment, all participants chose to receive ICBIT.
  Arms: Waiting List

SUMMARY:
To evaluate the effect and acceptability of an Internet-based comprehensive behavioral intervention for tics (ICBIT) in a sample of children and adolescents with Tic disorders. children and adolescents (aged 8-17 years) with Tourette Syndrome (TS) or Chronic Tic Disorder (CTD) and their parents will be randomly assigned to receive either an Internet-based ICBIT or wait-list (WL).

DETAILED DESCRIPTION:
To evaluate the effect and acceptability of an Internet-based comprehensive behavioral intervention for tics (ICBIT) in a sample of children and adolescents with Tic disorders, children and adolescents (aged 8-17 years) with Tourette Syndrome (TS) or Chronic Tic Disorder (CTD) and their parents will be randomly assigned to receive either an Internet-based ICBIT or wait-list (WL) condition in a cross over design.

Participants will be randomized to ICBIT, or to wait list, and half will cross over from wait list to ICBT. Two blind independent clinical evaluators will rate tic severity and comorbidity. The primary outcome measure is the Yale Global Tic Severity Scale (YGTSS). Assessments will be performed at baseline, post-ICBT or post wait list, 3-months and 6-months (post-treatment for those originally assigned to ICBT) and post-ICBT, 3-months and 6-months (post-treatment for those originally assigned to wait list condition). All assessments were conducted by 2 PhD level independent child psychologists.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Tourette Syndrome or Chronic Tic Disorder.
* Yale Global Tic Severity Scale tic severity score ≥14.

Exclusion Criteria:

* Change in psychotropic medication regimen during the past 6 weeks.
* Current diagnosis of substance abuse/dependence.
* Lifetime diagnosis of pervasive developmental disorder, mania or psychosis.
* Previous sessions of CBIT.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-01-31 (Estimated); Study Completion 2020-05-01 (Estimated)

PRIMARY OUTCOMES:
Yale Global Tic Severity Scale (YGTSS) | change from baseline YGTSS total score at 3 months

CONTACTS AND LOCATIONS:
Locations (2):
- Israel (2):
  - 1Interdisciplinary Center (IDC), Herzliya
  - Tel Aviv Sourasky Medical Center, Tel Aviv

REFERENCES:
- [Derived] Rachamim L, Zimmerman-Brenner S, Rachamim O, Mualem H, Zingboim N, Rotstein M. Internet-based guided self-help comprehensive behavioral intervention for tics (ICBIT) for youth with tic disorders: a feasibility and effectiveness study with 6 month-follow-up. Eur Child Adolesc Psychiatry. 2022 Feb;31(2):275-287. doi: 10.1007/s00787-020-01686-2. Epub 2020 Nov 24. PMID 33231786